CLINICAL TRIAL: NCT00904150
Title: A Case-control Study of the Molecular Genetics of Menstrual Migraine (Pure Menstrual and Menstrually-related Migraine)
Brief Title: Study of the Molecular Genetics of Menstrual Migraine
Status: Completed | Type: Observational
Sponsor: The City of London Migraine Clinic (Other)
Collaborators: Griffith University (Other)
Responsible Party: Principal Investigator, Dr E Anne MacGregor, Professor E Anne MacGregor, Queen Mary University of London
Other Study IDs: COLMC-GEN-2007; REC Ref: 07/H0703/107; Proposal # 36470; Grant Application 2007/03
Record Dates: First submitted 2009-05-17; First posted 2009-05-19 (Estimated); Results first posted 2014-02-24 (Estimated); Last update posted 2014-02-24 (Estimated); Status verified 2014-02

CONDITIONS: Migraine
Keywords: menstruation; migraine; menstrual migraine; genetics
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1 Menstrual migraine: Caucasian women with a current or past history of menstrual migraine (MM = pure menstrual migraine or menstrually-related migraine) attending the City of London Migraine Clinic
- 2 No migraine: Caucasian women with no personal history of migraine

SUMMARY:
The investigators hypothesize that genes that play a role in menstrual migraine can be identified using a well characterised migraine population and a comprehensive genome-wide association scan approach.

The aim of the study is to identify genes, genetic regions, and the effect of hormones on expression profiles in women with menstrual migraine compared to a control population with no personal or first-degree family history of migraine.

In this case control study, saliva samples will be taken from 300 cases and 300 controls for DNA analysis. Blood samples from 30 cases and 30 controls will be taken during the follicular phase as well as the luteal phase of the menstrual cycle for ribonucleic acid (RNA) analysis.

ELIGIBILITY:
Inclusion Criteria:

All cases and controls must:

* Be over 18 years
* Caucasian
* Provide written, informed consent
* Clearly understand and be able to comply with all the trial procedures, as required
* Not have taken part in trials of any investigational products within the previous 4 weeks

DNA Study:

* Cases must have at least a 12-month current or past history of menstrual migraine

RNA Study:

* Cases must have at least a 12-month current history of menstrual migraine
* Cases must have kept at least three months of headache diary data in advance of visit in order to confirm diagnosis
* Controls must still be having menstrual periods

Exclusion Criteria:

DNA Study:

* Cases and controls must not have smoked, chewed gum or consumed any food or drink in the 30 minutes prior to sample collection

RNA Study:

* Cases and controls will not be eligible for participation if they have:

  * Polycystic ovarian syndrome;
  * Taken any hormones or drugs in the previous three months that may affect normal hormone activity (e.g., hormonal contraceptives, hormone replacement therapy, dietary supplements such as isoflavones);
  * Donated or lost a significant amount of blood (> 550 mL) within the previous 12 weeks
  * Additionally, controls must not have a personal or family history in any first-degree relative of current or past migraine

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Caucasian women
Sampling Method: Non-Probability Sample
Enrollment: 585 (Actual)
Dates: Start 2007-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: E A MacGregor, FFSRH MD, Principal Investigator — Centre for Neuroscience and Trauma, Queen Mary, University of London; Lyn Griffiths, BSc(Hons) PhD, Principal Investigator — Genomics Research Centre Griffith University
Locations (1):
- The City of London Migraine Clinic, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Period: Saliva Samples (DNA)
Arm/Group | 1 Menstrual Migraine | 2 No Migraine
Started | 285 | 300
Completed | 282 | 155
Not Completed | 3 | 145
Not completed — saliva samples not suitable for assay | 3 | 0
Not completed — Australian samples of different genotype | 0 | 145
Period: Blood Samples (RNA): Follicular Phase
Arm/Group | 1 Menstrual Migraine | 2 No Migraine
Started | 37 | 32
Completed | 37 | 32
Not Completed | 0 | 0
Period: Blood Samples (RNA): Luteal Phase
Arm/Group | 1 Menstrual Migraine | 2 No Migraine
Started | 34 | 30
Completed | 34 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 1 Menstrual Migraine | 2 No Migraine | Total
Number analyzed (Participants) | 285 | 300 | 585
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 285 | 300 | 585
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 285 | 300 | 585
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United Kingdom | 285 | 155 | 440
  Australia | 0 | 145 | 145

OUTCOME MEASURES:

1. Primary Outcome: Progesterone Receptor Gene Polymorphism PROGINS in Women With Menstrual Migraine and Women Without Migraine
Description: PR PROGINS
Time Frame: 6 years
Population: Not all samples were suitable for analysis for each outcome measure
Measure: Number; unit: participants
Arm/Group | 1 Menstrual Migraine | 2 No Migraine
Number analyzed (Participants) | 280 | 153
participants
  No PROGINS insert | 208 | 112
  Heterozygote | 64 | 39
  Homozygote | 8 | 2
Statistical Analysis 1: Comparison: 1 Menstrual Migraine vs 2 No Migraine; Statistical analysis is of the distribution of PR PROGINS polymorphism frequencies between groups; Test type: Superiority or Other; p = 0.513, Chi-squared

2. Primary Outcome: Estrogen Receptor 1 G594a Polymorphism in Women With Menstrual Migraine and Women Without Migraine
Description: ESR1 G594A
Time Frame: 6 years
Population: Not all samples were suitable for analysis for each outcome measure
Measure: Number; unit: participants
Arm/Group | 1 Menstrual Migraine | 2 No Migraine
Number analyzed (Participants) | 280 | 150
participants
  Genotype GG | 196 | 101
  Genotype GA | 76 | 43
  Genotype AA | 8 | 6
Statistical Analysis 1: Comparison: 1 Menstrual Migraine vs 2 No Migraine; Statistical analysis is of the distribution of Estrogen receptor 1 G594a polymorphism frequencies between groups; Test type: Superiority or Other; p = 0.75, Chi-squared

3. Secondary Outcome: Tumour Necrosis Factor Genotype in Women With Menstrual Migraine and Women Without Migraine
Description: TNF
Time Frame: 6 years
Population: Not all samples were suitable for analysis for each outcome measure
Measure: Number; unit: participants
Arm/Group | 1 Menstrual Migraine | 2 No Migraine
Number analyzed (Participants) | 190 | 54
participants
  Genotype GG | 1 | 2
  Genotype GA | 40 | 20
  Genotype AA | 149 | 32
Statistical Analysis 1: Comparison: 1 Menstrual Migraine vs 2 No Migraine; Analysis of distribution of TNF genotype frequencies between groups; Test type: Superiority or Other; p = 0.002743, Chi-squared; Odds Ratio (OR) = 0.434, 95% CI [0.24 to 0.75]

4. Secondary Outcome: SYNE1 Genotype in Women With Menstrual Migraine and Women Without Migraine
Description: SYNE1
Time Frame: 6 years
Population: Not all samples were suitable for analysis for each outcome measure
Measure: Number; unit: participants
Arm/Group | 1 Menstrual Migraine | 2 No Migraine
Number analyzed (Participants) | 215 | 119
participants
  Genotype TT | 24 | 25
  Genotype TG | 102 | 54
  Genotype GG | 89 | 40
Statistical Analysis 1: Comparison: 1 Menstrual Migraine vs 2 No Migraine; Analysis of distribution of SYNE1 genotype frequencies between groups; Test type: Superiority or Other; p = 0.02462, Chi-squared; Odds Ratio (OR) = 0.69, 95% CI [0.49 to 0.95]

5. Primary Outcome: Estrogen Receptor 1 C325G Polymorphism in Women With Menstrual Migraine and Women Without Migraine
Description: ESR1 C325G
Time Frame: 6 years
Population: Not all samples were suitable for analysis for each outcome measure
Measure: Number; unit: participants
Arm/Group | 1 Menstrual Migraine | 2 No Migraine
Number analyzed (Participants) | 280 | 154
participants
  Genotype CC | 155 | 96
  Genotype CG | 109 | 51
  Genotype GG | 16 | 7
Statistical Analysis 1: Comparison: 1 Menstrual Migraine vs 2 No Migraine; Statistical analysis is of the distribution of Estrogen receptor 1 C325G polymorphism frequencies between groups; Test type: Superiority or Other; p = 0.18, Chi-squared

6. Primary Outcome: Menstrual Cycle Expression of PGR and ESR in Women With Menstrual Migraine and Women Without Migraine
Description: PgR and ESR
Time Frame: 6 years
Population: Matched pairs of follicular and luteal samples Not all samples were suitable for analysis for each outcome measure
Measure: Mean (Standard Deviation); unit: number of genes expressed
Arm/Group | 1 Menstrual Migraine | 2 No Migraine
Number analyzed (Participants) | 30 | 29
number of genes expressed
  ESR expression in follicular phase | 15.98 (NA) — Data not reported | 16.73 (NA) — Data not reported
  ESR expression in luteal phase | 16.58 (NA) — Data not reported | 15.62 (NA) — Data not reported
  PGR expression in follicular phase | 9.62 (NA) — Data not reported | 9.80 (NA) — Data not reported
  PGR expression in luteal phase | 8.95 (NA) — Data not reported | 8.69 (NA) — Data not reported
Statistical Analysis 1: Comparison: 1 Menstrual Migraine vs 2 No Migraine; Test type: Superiority or Other; p > 0.05, t-test, 1 sided

7. Secondary Outcome: Menstrual Cycle Expression of TNF and SYNE1 in Women With Menstrual Migraine and Women Without Migraine
Description: TNF and SYNE1
Time Frame: 6 years
Population: Matched luteal and follicular phase samples Not all samples were suitable for analysis for each outcome measure
Measure: Mean (Standard Deviation); unit: number of genes expressed
Arm/Group | 1 Menstrual Migraine | 2 No Migraine
Number analyzed (Participants) | 29 | 29
number of genes expressed
  TNF expression in follicular phase | 17.16 (NA) — Not reported | 17.33 (NA) — Not reported
  TNF expression in luteal phase | 16.24 (NA) — Not reported | 16.96 (NA) — Not reported
  SYNE1 expression in follicular phase | 21.56 (NA) — Not reported | 20.68 (NA) — Not reported
  SYNE1 expression in luteal phase | 20.01 (NA) — Not reported | 20.06 (NA) — Not reported
Statistical Analysis 1: Comparison: 1 Menstrual Migraine vs 2 No Migraine; Test type: Superiority or Other; p > 0.05, t-test, 1 sided

ADVERSE EVENTS:
Description: This is not an interventional study so serious and another [non-serious] adverse events could not be assessed.
Arm/Group | 1 Menstrual Migraine | 2 No Migraine
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No